

# Wise Intervention for the Reduction of Aggressive Behaviors and the Promotion of Prosocial Behaviors toward LGB-TNB People

**Informed consent** 

**September 25, 2025** 

University of Deusto. Bilbao.



# FACULTY OF HEALTH SCIENCES/ UNIVERSITY OF DEUSTO

#### Dear Family,

From the Deusto Stress Research team, we would like to introduce you to a research project currently being carried out at the University of Deusto. The aim of this project is **to examine the effects of two brief school-based interventions on reducing aggressive behaviors and promoting prosocial behaviors in both virtual and face-to-face settings, as well as on improving adolescents' healthy habits. This is especially important because adolescence is a developmental stage in which new experiences are common, which can sometimes lead to engagement in risky behaviors. In addition, during this stage, discrimination and aggression among peers increase, with certain groups being particularly vulnerable (e.g., LGBT individuals, neurodivergent individuals, etc.). Although the visibility of diversity has increased in recent years, aggression toward minority groups continues to occur at a higher rate than in other sectors of the population.** 

Below you will find all the relevant information regarding the project. Once you have read the information, if you do **NOT** want your son/daughter to participate in this project, please fill out the consent form and return it to your child's school within 3 days. If you authorize your son/daughter to participate, you do not need to complete the form or return it.

#### **Purpose of the Project**

The aim of this project is to evaluate the effectiveness of two formats of brief smart interventions: one focused on reducing aggressive behaviors and promoting prosocial behaviors among peers, and the other on fostering healthy habits in adolescents. Therefore, the interventions aim to (1) reduce aggressive behaviors among peers, (2) promote prosocial behaviors, and (3) improve healthy habits.

The intervention will take place in a single session lasting approximately 60 minutes. Two intervention formats will be used, with adolescents randomly assigned to each of them. Afterwards, all participants will have the opportunity to receive the other intervention format if it proves to be effective.

The interventions consist of completing exercises such as: (1) reading scientific information about social behavior and its role in people's well-being, (2) reading, reflecting, and writing about the meaning and value of prosocial and aggressive behaviors through stories and experiences of their own and of other young people their age, and (3) self-persuasion exercises that involve an active commitment to change. All students in your son/daughter's class have received the invitation to participate.

We believe that this project **has significant potential to improve coexistence** among students.

#### Who is it aimed at?

Several schools **in Bizkaia and Cantabria** have received the invitation to participate, and it is estimated that up to a total of 1,000 students between the ages of 14 and 18 will take part in the study.

#### What will your son/daughter be asked to do?

If you allow your son/daughter to take part in this study, he/she will be asked to

- Participate in the intervention and subsequent evaluation lasting 60 minutes.
- Complete a questionnaire of about 50 minutes one week before the intervention, and three, six, and nine months after the intervention.

#### How will the researchers protect the privacy of the participants?

The study will be carried out with the support of the Basque Government and has been approved by the Research Ethics Committee of the University of Deusto [Ref: ETK-90/24-25]. The researchers will protect the privacy of all participants. Participation is anonymous, so no first or last names will be indicated anywhere. The evaluation and intervention data will be linked through a code known only to the participants.

#### How will the researchers share the results of the project?

Your son/daughter's school will receive a final report that will reflect the results of the program evaluation and may be distributed to all families.

## Are there any risks or benefits for my son/daughter?

Participation in this study does not involve physical risks, but there is a possibility that some participants may experience emotional discomfort when responding to the battery of questionnaires or during the intervention. If this occurs, the research team will provide support and reassurance. In addition, participants will be offered the option to complete an alternative activity or withdraw from the study if they wish, without any negative consequences. Furthermore, all participants will be provided with relevant contact information for their well-being, including helpline numbers for children and adolescents and the email address of the principal investigator of the project, who will be available for any questions or requests for support after participation. Likewise, conducting this study may contribute to the reduction of aggressive and discriminatory behaviors among students, while promoting prosocial and supportive behaviors when witnessing aggressive behaviors.

#### Is my son/daughter required to participate?

Consent and participation are **voluntary**. Families will have to decide whether their son/daughter participates in the study. The decision to allow or not allow your son/daughter to participate will not affect the relationship with the school or with the University of Deusto. In addition to the families' permission, your son/daughter must also agree to participate in the study. If they do not wish to participate, they will not be included in the study and there will be no penalty. Even if both the family and your son/daughter initially agree to participate in the study, you may change your mind later without any type of penalty.

This project will be carried out during the regular classroom activities. However, if you do not want your son/daughter to participate, a different activity will be available. They will be given the option to use their time to read or to do schoolwork.

#### Will there be any compensation?

There will be no monetary compensation for participating. However, as a token of appreciation for the effort made, those who take part in the study will be entered into a raffle for several **gift vouchers** to be used in department stores. The raffle will be held at the time of the final data collection.

## Who has reviewed the study?

The project has been reviewed by the Ethics Committee of the University of Deusto and by the management of the schools. The school will not carry out the project activities. The study will be conducted by researchers from the University of Deusto.

# Who can I contact if I have questions about the project?

Before, during, or after participation in the project, you may contact any of the following people:

[Masked]

# This document should only be signed if you do **NOT** want your daughter/son to participate in the project.

I agree with the conditions specified above and understand that I can withdraw my daughter/son from the project at any time and that my daughter/son may choose not to answer any of the questions if she/he does not wish to answer them. I understand that my daughter/son's participation is completely voluntary, confidential, and anonymous.

Your signature indicates that you have read the information and have decided **NOT** to allow your daughter/son to participate in this project. <u>If you give your permission for your daughter/son to participate, you do not need to complete this form.</u>

□ NO, my daughter/son may NOT participate in the project

Full name of your daughter/son:

Signature of mother, father, or legal guardian:

Date